CLINICAL TRIAL: NCT01842399
Title: Resveratrol and Cardiovascular Health in the Elderly: The Reache Trial
Brief Title: Resveratrol and Cardiovascular Health in the Elderly
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The protocol experienced slow accrual.
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 130078; 13-AG-0078
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Vascular Resistance; Hypertension
Keywords: Vascular Stiffness; Aging; Resveratrol; Aerobic Capacity; Inflammation
MeSH Terms: conditions — Hypertension; Inflammation | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Comparator (Placebo Comparator): 2x/day orally
  Interventions: Drug: Placebo
- Resveratrol 1 (Experimental): 75 mg, 2x/day orally
  Interventions: Dietary Supplement: Resveratrol
- Resveratrol 2 (Experimental): 150 mg, 2x/day orally
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — Nutriceutical
  Arms: Resveratrol 1; Resveratrol 2
Drug: Placebo — 2x/day orally
  Arms: Placebo Comparator

SUMMARY:
Background:

- Resveratrol is a compound found in the skin of red grapes. It is being tested to see if it can have positive effects on human health. Lab studies show that it may help lower blood sugar, improve heart and blood vessel health, and prevent cancer. Researchers want to test different dose levels of Resveratrol to see what kind of effects it has on older overweight people. It will be tested in healthy volunteers at least 50 years of age.

Objectives:

- To test the effects of different dose levels of Resveratrol on heart and blood vessel health.

Eligibility:

- Healthy overweight nonsmoking volunteers at least 50 years of age.

Design:

* This study will involve a screening visit and four study visits. Some of the study visits will involve overnight inpatient stays.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. They will be given a list of foods that they should avoid eating while on the study.
* Participants will be separated into three groups. Two groups will take different dose levels of the study drug. The third group will take a placebo.
* At the first study visit, participants will stay in the clinical center overnight for 2 days of tests. They will provide blood and urine samples and have body scans to measure fat and muscle mass. They will also have exercise tests. A muscle biopsy will also be performed. At this visit, they will receive their dose of the study drug. They will continue to take this dose for as long as they are on the study.
* The second visit will be 16 weeks after the first one. It will take only 2 hours, and repeat most of the tests from the screening visit.
* The third visit will be 16 weeks later. It will involve an overnight stay. Most of the tests from the second visit will be repeated.
* The fourth and final visit will be 16 weeks later. It will involve an overnight stay. Most of the tests from the initial study visit (including the scans and the exercise tests) will be repeated.

DETAILED DESCRIPTION:
Resveratrol is found in the leaves and skin of grapes, in peanuts and in the roots of the plant polygonum cupsidatum. Although used since early years in Indian Ayurvedic and Chinese medicine, it came into prominence in the 1990 s as it was believed to be the major reason for the positive effect of wine on cardiovascular health and the French Paradox. Since then, studies have shown that resveratrol affects a number of key cellular pathways and molecular targets with a wide range of biological effects. Noted among these are its effects on the blood vessels, cancer, blood clotting, blood sugar control, cognition, muscle activity and inflammation. Resveratrol also may produce some of the same effects as decreased food intake, perhaps through its action on a molecule in the body called Sirtuin, which is important because this is one of the only approaches that has consistently demonstrated beneficial effects on the aging process.

Resveratrol s action and pharmacology has been extensively studied in test tubes, cells, and animals but is only now being explored fully in people. The animal studies include a recent NIA-conducted study in monkeys that demonstrated a reduction in the stiffness of blood vessel over several weeks. Phase 1 and 2 clinical studies in healthy human volunteers or in patients with type II diabetes mellitus have begun to identify possible roles for resveratrol as a dietary supplement and the compound appears to have no harmful effects at doses up to 5 grams per day. There is also growing interest in pharmacological interventions targeting cardiovascular risk factors such as atherosclerosis and type II diabetes to prevent neurodegenerative diseases such as Alzheimer s disease (AD).

We will perform a 12-month trial of resVida (an oral preparation of resveratrol) in 120 randomized overweight/obese people over the age of 50 (40 in each group). This is a Phase 1 and 2 double-blind randomized study. One of two doses of study compound (75mg twice daily or 150mg twice daily) or placebo will be self-administered twice a day for 52 weeks to participants 50 years or older. The primary endpoint will be vascular stiffness (as measured by Pulse Wave Velocity) and the secondary endpoint will be exercise capacity as measured by oxygen utilization (VO2max). Testing will be done on the levels of resveratrol in the blood with different doses of the compound. The study will also include measurements of changes in blood glucose levels, inflammation, and exercise capacity. Targeted, quantitative metabolomics assays in blood will be performed to test whether concentrations of small metabolites previously shown to be associated with arterial stiffness, including free oxysterols, amino acids, acycarnitines and glycerophospholipids are modulated by resveratrol. These studies will provide necessary information for further testing of resVida as a compound that could promote healthy aging.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male or Female, age 50 years or older

BMI greater than or equal to 25 or less than or equal to 35 and weight less than 300 pounds.

Participants must provide their own consent.

Females must be menopausal or have had a bilateral oophorectomy.

* If over 55 years old: no menses for 12 months or longer. Women over 55 years old who haven't had a period for a year will be considered menopausal and do not need a FSH test.
* If 50-55 years old: no menses for 12 months AND an FSH level greater than or equal to 20. Women between 50 and 55 years old who haven't had a period for a year, will need FSH test. If their FSH test is more than 20, they will be considered menopausal. If their FSH test is less than 20, they will not be eligible to participate.

EXCLUSION CRITERIA:

Liver Function Tests (LFT) greater than 2 times normal.

Abnormal thyroid function, as evidenced by Free T3, t4, Free T4 or TSH +/- 5% of the lab reference ranges

History of diabetes (gestational diabetes ok).

Hemoglobin A1C greater than 6.5 and/or fasating serum glucose greater than or equal to 126 mg/dL.

Renal dysfunction (GFR less than 60 mL/min).

Abnormal Coagulation profile (PT/PTT and INR).

Medications: (Due to potential interaction with resveratrol)

Cholesterol medications Atorvastatin(Lipitor) Rosuvastatin (Crestor), Simvastatin (Zocor), Gemfibrazole (Lopid), Niacin (Niacor), etc.

Aspirin greater than 81 mg

* Taking medicines that may increase the risk of bleeding such as Coumadin (warfarin), Plavix (clopidogrel), Xarelto (rivaroxaban), Pradaxa (dabgatran), Eliquis (apixaban) or Heparin (blood thinning medications) due to their potential interaction with resveratrol and the increased risk for bleeding with the muscle biopsy.
* Taking supplements such as Ginkgo biloba, Ginseng or Ginger due to their increased risk of bleeding with the muscle biopsy.
* Chronic (daily) use of non-steroidal anti-inflammatory agents (NSAIDs) such as Motrin (Ibuprofen), Advil (Ibuprofen) or Naprosyn (Naproxen)-due to potential interaction with resveratrol. (Occasional use is ok if the participant does not take them 4 days before and 3 days after the muscle biopsy procedure).

Anti-diabetic medications: Insulin, Metformin (Glucophage, Avandamet, Glibomet, etc), Rosiglitazone (Avandia), Exenatide (Byetta), Sitagliptin (Januvia), etc

Testosterone and estrogen supplement

Current glucocorticoid use, or up to 3 months ago (nasal, topical, ophthalmic, and inhaled use are not exclusionary)

Vitamin supplements containing resveratrol

Contraindications to MRI Study; e.g. metal implants, pacemakers, etc and hip replacements (metal or plastic) due to inhibiting visualization of the area being scanned.

Smoking nicotine presently or within the last 3 months.

Known congestive heart failure now or in the past.

Alcohol consumption more than 30 grams (equivalent to about 10 ounces of wine; 24 ounces of beer; 3 ounces of hard liquor) for men or 15 grams for women (equivalent to about 5 ounces of wine; 12 ounces of beer; 1.5 ounces of hard liquor) daily.

Positive screening result for alcohol use at the screening visit. Score 8+ on the AUDIT.

Positive HIV, Hepatitis B or C testing.

Positive urine drug test (exclusionary due to unknown interaction affect with study medication and question of compliance with study procedures).

* Benzodiazepines
* Amphetamines
* Barbiturates
* Cannabis
* Cocaine

Receipt of any investigational products (e.g. drugs, supplements, dietary interventions) as part of a research study within 30 days of initial dose administration

Unable to comply with the study requirements and procedures.

Unable to perform treadmill testing due to reasons such as orthopedic problems, moderate to severe aortic stenosis as found on echocardiogram at ScreeningVisit, history of myocardial infarction in the last three months or angina (under treatment).

Unable to perform knee strength testing due to reasons such as bilateral knee replacements.

Unable to perform hand grip testing due to any limitation such as pain or deformity.

Allergy or intolerance to local anesthetic- Lidocaine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
To determine if oral resveratrol administered for 12 months will blunt the aging associated increase in vascular stiffness as measured by Pulse Wave Velocity (PWV). | Week 16, 32, 52
  Decreased rate of age associated arterial stiffening

SECONDARY OUTCOMES:
To determine if oral resveratrol administered for 12 months will improve exercise capacity as measured by MVO2-treadmill. | Week 16, 32, 52
  Changes in aerobic capacity, functional capacity, body composition, muscle energetics, inflammatory markers, glucose metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Ajoy C Karikkineth, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-AG-0078.html